CLINICAL TRIAL: NCT01807104
Title: Prospective Randomized Single Center Clinical Evaluation of THA Surgical Techniques Comparing the Direct Anterior Approach to the Posterior Approach
Brief Title: Total Hip Arthroplasty (THA) Surgical Techniques Comparing the Direct Anterior Approach to the Posterior Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barrett, William, M.D. (Individual)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, William Barrett, M.D., William Barrett,M.D,, Barrett, William, M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20091819
Record Dates: First submitted 2011-06-16; First posted 2013-03-08 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-07

CONDITIONS: Osteoarthritis of the Hip
Keywords: Anterior Approach; Posterior Approach
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anterior Approach Total Hip (Active Comparator): Total hip arthroplasty performed through an anterior surgical approach. Compare results of total hip arthroplasty performed through either an Anterior or Posterior Surgical Approach
  Interventions: Procedure: Anterior Approach / Posterior Approach
- Posterior Approach Total Hip (Active Comparator): The additional arm is the posterior approach total hip, which the Anterior Approach is being compared too. Compare results of total hip arthroplasty performed through either an Anterior or Posterior Surgical Approach.
  Interventions: Procedure: Anterior versus Posterior Approach for total hip replacement

INTERVENTIONS:
Procedure: Anterior Approach / Posterior Approach — compare results of total hip arthroplasty performed through either an anterior or posterior surgical approach
  Arms: Anterior Approach Total Hip
Procedure: Anterior versus Posterior Approach for total hip replacement — Compare results of total hip arthroplasty performed through either an anterior or posterior surgical approach
  Arms: Posterior Approach Total Hip

SUMMARY:
The purpose of this study is to compare the short term effectiveness and return to function of subjects undergoing primary Total Hip Arthroplasty using an Anterior Approach (incision on the front part of the hip joint) versus Posterior Approach (incision over back part of the hip joint).

DETAILED DESCRIPTION:
The anterior approach may provide better early post-operative outcomes because there are fewer muscles at the front of the hip so the surgeon works between them rather than cutting through muscle fibers. However, the anterior approach is more difficult to access so usually requires a specialized table.

The posterior approach is easier to access, but the incision cuts through muscle fiber. This may lengthen recovery time. However, a specialized table, which can be quite expensive, is often not required.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to or capable of providing consent to participate in the clinical investigation.
2. Subject is between the ages of 20-75 years, inclusive.
3. Subject requires a cementless, primary total hip arthroplasty for non-inflammatory degenerative joint disease (NIDJD)
4. Subject has sufficient bone stock for the hip replacement device.
5. Subject is a suitable candidate for the devices specified in the clinical investigation plan and is willing to be randomized to either surgical approach.

Exclusion Criteria:

1. Subject in the opinion of the Investigator has an existing condition that would compromise his /her participation and follow-up in this investigation.
2. Subject has had previous surgery on the affected hip.
3. Subject has significant osteoarthritis of the contra-lateral hip requiring a total hip arthroplasty within 12 months.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P Barrett, MD, Principal Investigator
Locations (1):
- Valley Orthopedic Associates, Renton, Washington, United States

REFERENCES:
- See also: Prospective, Randomized Study of Direct Anterior Approach vs Posterolateral Approach Total Hip Arthroplasty: A Concise 5-Year Follow-Up Evaluation — https://doi.org/10.1016/j.arth.2019.01.060

RESULTS

PARTICIPANT FLOW:
Groups:
- Direct Anterior Approach: Direct Anterior Approach (DAA) utilizing a modern fracture table with the patient placed supine, both feet in boots for proper positioning. Anterior skin incision, 10-14 cm long, is used. An inter-muscular plane is utilized to access the anterior hip capsule. The hip capsule is opened anteriorly, a femoral neck osteotomy is performed based on pre-operative templating, and the femoral head removed. Acetabular retractors are placed and reaming of the acetabulum commenced. This is done under direct visualization with C-arm confirmation for positioning. The femoral side is then visualized with the aid of the fracture table. A hydraulic trochanteric hook elevates the proximal femur. Broaching of the femoral canal is started and proceeds up to the appropriate size. A trial reduction is performed, and the length and offset are checked manually and with C-arm confirmation. The trial components are removed and the prostheses are placed with press-fit fixation. Routine closure is performed.
- Postero-Lateral Approach: Postero-Lateral Approach (PA) uses a standard OR table with the patient placed in the lateral decubitus position. A 10-14 cm skin incision is utilized over the posterior-lateral corner of the hip. The gluteus maximus muscle is split in line with its fibers and the short external rotators and posterior capsule are opened. The hip is dislocated posteriorly and a femoral neck osteotomy is performed. The acetabular and femoral components are inserted in the same manner as is done with the DAA with press fit fixation utilized. The PA is well described in all major texts on orthopedic surgery.
Period: Overall Study
Arm/Group | Direct Anterior Approach | Postero-Lateral Approach
Started | 43 | 44
Completed | 39 | 40
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Anterior Approach | Postero-Lateral Approach | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (9.0) | 63.0 (8.0) | 62.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 25 | 39
  Male | 29 | 19 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 43 | 44 | 87
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Returning to Quality of Life by Using Either Anterior Approach Versus Posterior Approach
Description: Harris Hip 5-Year Total Score Change from Baseline. The Harris Hip score gives a maximum of 100 points. Pain receives 44 points, function 47 points, range of motion 5 points, and deformity 4 points. Function is subdivided into activities of daily living (14 points) and gait (33 points). The higher the Harris Hip score, the less dysfunction.This outcome measure has been validated for joint replacement surgery for peer reviewed orthopedic literature.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Direct Anterior Approach | Postero-Lateral Approach
Number analyzed (Participants) | 38 | 40
score on a scale | 40.1 (10.89) | 43.8 (15.94)

ADVERSE EVENTS:
Time Frame: 8 years
Arm/Group | Direct Anterior Approach | Postero-Lateral Approach
All-Cause Mortality (participants affected / at risk) | 1/43 | 1/44
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44
Other Adverse Events (participants affected / at risk) | 5/43 | 6/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Direct Anterior Approach (N=43) | Postero-Lateral Approach (N=44)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-01-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT01807104/Prot_SAP_000.pdf